CLINICAL TRIAL: NCT05926024
Title: Long-Term Follow-Up in Women With Early Breast Cancer Three Years of More Post Primary Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2229
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Quality of life; Adverse Events; Cancer free
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Women who participated in previous studies namely NCT02167932, NCT02328313, and NCT03761706, will be re-contacted and consented to study activities.
  Interventions: Diagnostic Test: p16 tumor suppressor gene
- Cohort B: Women with breast cancer, who did not receive chemotherapy, will be consented to be included in the study, and their electronic medical data will be used.
  Interventions: Behavioral: Exercise Recall Patient Reported Outcomes; Behavioral: Health Behavior Questionnaire (HBQ)30 Patient Reported Outcomes; Behavioral: Functional Assessment of Cancer Therapy-General (FACT-G) Patient Reported Outcomes; Behavioral: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Patient Reported Outcomes; Behavioral: Patient Reported Outcomes PROMIS Cognitive Function (Short Form 8a); Behavioral: Patient Reported Outcomes Functional Assessment of Cancer-Gynecology Oncology Group-Neurotoxicity (FACT/GOG-NTX-12); Behavioral: Patient Reported Outcomes PROMIS; Behavioral: Patient Reported Outcomes FACT-Endocrine Symptoms; Behavioral: Patient Reported Outcomes Penn Arthralgia Aging Survey; Behavioral: Patient Reported Outcomes PRO-CTCAE (patient-reported CTCAE); Diagnostic Test: p16 tumor suppressor gene

INTERVENTIONS:
Behavioral: Exercise Recall Patient Reported Outcomes — Questionnaire items inquire about (1) the number of days of the week participants engage in walking for pleasure or exercise and (2) the number of minutes per day that participants engage in walking for pleasure or exercise. The same two questions are repeated pertaining to exercise in general. Completion of these items takes 1 minute to complete.
  Groups: Cohort B
Behavioral: Health Behavior Questionnaire (HBQ)30 Patient Reported Outcomes — Health Behavior Questionnaire (HBQ)30 -- Questionnaire items pertain to the history of smoking, engagement in vigorous physical activity, alcohol consumption, and mortality status of parents, and take less than 1 minute to complete.
  Groups: Cohort B
Behavioral: Functional Assessment of Cancer Therapy-General (FACT-G) Patient Reported Outcomes — Functional Assessment of Cancer Therapy-General (FACT-G) is a quality of life and function measure developed and validated over 20 years ago that has been used in hundreds of cancer studies worldwide. It consists of four well-being domains -- physical, social/family, emotional, and functional. The FACT-G (Version 4) is a 27-item instrument that is formatted for self-administration and uses a 5-point Likert-type scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). The recall period is "during the past 7 days". It takes 6-8 minutes for an average patient to complete.
  Groups: Cohort B
Behavioral: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Patient Reported Outcomes — Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) is a 13-item scale that uses a 5-point Likert-type scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). The recall period is "during the past 7 days". This measure takes about 1 minute to complete.
  Groups: Cohort B
Behavioral: Patient Reported Outcomes PROMIS Cognitive Function (Short Form 8a) — PROMIS Cognitive Function (Short Form 8a) includes 8 items on a 5-point Likert-type scale ranging from very often/several times a day = 1 to never = 5, with higher scores indicating greater perceived loss of cognitive function. This measure takes less than 1 minute to complete.
  Groups: Cohort B
Behavioral: Patient Reported Outcomes Functional Assessment of Cancer-Gynecology Oncology Group-Neurotoxicity (FACT/GOG-NTX-12) — Functional Assessment of Cancer-Gynecology Oncology Group-Neurotoxicity (FACT/GOG-NTX-12) is a questionnaire that includes 12 items inquiring about symptoms in the past 7 days (0=not at all to 4=very much) pertaining to numbness or tingling in hands/feet, discomfort in hands/feet, joint pain or muscle cramps, weakness all over, trouble hearing, ringing/buzzing in ears, buttoning buttons, trouble feeling the shape of small objects in hands, trouble walking, and pain in hands/feet in cold temperatures. This measure takes about t 1 minute to complete.
  Groups: Cohort B
Behavioral: Patient Reported Outcomes PROMIS — PROMIS Measures Global Health (10 items), Anxiety (6 items), Depression (8 items), and Stress (10 items). All items are on a 5-point Likert-type scale form never to very often. Completion of all 34 items should take no more than 3 minutes to complete.
  Groups: Cohort B
Behavioral: Patient Reported Outcomes FACT-Endocrine Symptoms — FACT-Endocrine Symptom is a 19-item questionnaire inquiring about hot flashes, cold sweats, night sweats; vaginal discharge, itching/irritation, bleeding or spotting, dryness; pain or discomfort with intercourse, loss of interest in sex; weight gain; lightheadedness; vomiting; diarrhea; headaches; bloating; breast sensitivity/tenderness; mood swings; irritability; pain in joints. Responses are on a 5- point Likert-type scale from not at all to very much. This measure takes about two minutes to complete.
  Groups: Cohort B
Behavioral: Patient Reported Outcomes Penn Arthralgia Aging Survey — Penn Arthralgia Aging Survey is an 8-item scale inquiring about joint pain, with a 4-point response scale from not at all to complete. Items pertaining to slowing down, stopping, being hesitant, unable to do this, and feeling unusually aged. This measure takes less than a minute to complete.
  Groups: Cohort B
Behavioral: Patient Reported Outcomes PRO-CTCAE (patient-reported CTCAE) — PRO-CTCAE (patient-reported CTCAE) is Patients will be asked about the side effects of chemotherapy treatment at baseline, every 3 weeks during chemotherapy, at the end of chemotherapy, and at 6 months post-chemotherapy. Patients are asked to rate "in the past 7 days" the average severity, frequency, and intensity and a scale from 1=none/never/not at all to 5=very severe/very much/almost all of the time. Symptom list: Abdominal pain, Constipation, Diarrhea. Mucositis oral, Nausea, Vomiting, Edema limbs, Fatigue, Pain, Arthralgia, Myalgia, Peripheral sensory neuropathy, Anxiety, Depression, Insomnia, Dyspnea, Rash maculopapular, Hot flashes. Completion of these measures takes 5 minutes for an average patient
  Groups: Cohort B
Diagnostic Test: p16 tumor suppressor gene — Blood samples will be obtained to test the p16 tumor suppressor gene from the subjects It is voluntary..

SUMMARY:
This study evaluates whether there are pre-treatment factors such as patient characteristics, specific breast cancer type, specific treatments, toxicities, or adverse events during treatment that may impact the quality of life and function, 3 years or more after the treatment, in cancer-free subjects.

There will be 2 groups. Cohort A: Women who participated in previous studies namely NCT02167932, NCT02328313, and NCT03761706, will be re-contacted and consent for this study activities. Cohort B: Women with breast cancer, who did not receive chemotherapy, will be consented to be included in the study, and their electronic medical data will be used.

Furthermore, the long-term effects of treatment and a biomarker of aging cyclin-dependent kinase inhibitor 2A (CDKN2A,p16INK4a) and relation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

1. Informed consent was obtained per Institutional Review Board guidelines to participate in the study and HIPAA authorization for the release of personal health information.
2. Subjects are willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.
3. Age ≥21 years at the time of consent.
4. Able to read and comprehend English.
5. No breast cancer recurrence or metastasis; no other cancer diagnosis other than basal cell or squamous cell cancers.

Exclusion Criteria:

1. Unable to read or comprehend English.
2. Breast cancer recurrence or metastasis; any other cancer diagnosis other than basal cell or squamous cell cancer.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women have been diagnosed with breast cancer and cancer-free for equal or more than 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Well-being | At least 3 years after completion of chemotherapy
  Change in Functional Well-being will be measured by FACT-G Functional Well-bein in participants who received chemotherapy (Cohort A).
  Functional Assessment of Cancer Therapy-General (FACT-G) is a quality of life and function measure developed and validated over 20 years ago that has been used in hundreds of cancer studies worldwide. It consists of four well-being domains -- physical, social/family, emotional, and functional. The FACT-G (Version 4) is a 27-item instrument that is formatted for self-administration and uses a 5-point Likert-type scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). The recall period is "during the past 7 days". It takes 6-8 minutes for an average patient to complete.

SECONDARY OUTCOMES:
Comparison of Functional well-being- Cohort B | At least 3 years after completion of chemotherapy
  Comparison of Functional well-being will be measured as a comparison of FACT-G Functional Well-being scores of participants who received chemotherapy (Cohort A)and participant who did not receive chemotherapy (Cohort B).
  Functional Assessment of Cancer Therapy-General (FACT-G) is a quality of life and function measure developed and validated over 20 years ago that has been used in hundreds of cancer studies worldwide. It consists of four well-being domains -- physical, social/family, emotional, and functional. The FACT-G (Version 4) is a 27-item instrument that is formatted for self-administration and uses a 5-point Likert-type scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). The recall period is "during the past 7 days". It takes 6-8 minutes for an average patient to complete.
Changes in self-reported cognition-Cohort A | Pre-chemotherapy and at least 3 years after completion of chemotherapy
  Changes in self-reported cognition will be assessed using PROMIS Cognitive Function (Short Form 8a), between pre-chemotherapy and at least 3 years after completion of chemotherapy in the Cohort A group (participants who received chemotherapy).
  PROMIS Cognitive Function (Short Form 8a) This measure includes 8 items on a 5-point Likert-type scale ranging from very often/several times a day = 1 to never = 5, with higher scores indicating greater perceived loss of cognitive function.
Changes in self-reported cognition- Cohort B | Pre-chemotherapy and at least 3 years after completion of chemotherapy
  Changes in self-reported cognition will be assessed using PROMIS Cognitive Function (Short Form 8a), between pre-chemotherapy and at least 3 years after completion of chemotherapy in the Cohort B group (participants did not receive chemotherapy).
  PROMIS Cognitive Function (Short Form 8a) This measure includes 8 items on a 5-point Likert-type scale ranging from very often/several times a day = 1 to never = 5, with higher scores indicating greater perceived loss of cognitive function.
Changes in self-reported peripheral neuropathy-Cohort A | Pre-chemotherapy and at least 3 years after completion of chemotherapy
  Changes in self-reported peripheral neuropathy will be assessed using Functional Assessment of Cancer-Gynecology Oncology Group-Neurotoxicity (FACT/GOG-NTX-12), between pre-chemotherapy and at least 3 years after completion of chemotherapy in the Cohort A group (participants who received chemotherapy).
  FACT/GOG-NTX-12 is a questionnaire that includes 12 items inquiring about symptoms in the past 7 days (0=not at all to 4=very much) pertaining to numbness or tingling in hands/feet, discomfort in hands/feet, joint pain or muscle cramps, weakness all over, trouble hearing, ringing/buzzing in ears, buttoning buttons, trouble feeling the shape of small objects in hands, trouble walking, and pain in hands/feet in cold temperatures. The increasing score reflects worse neuropathy.
Changes in self-reported peripheral neuropathy-Cohort B | Pre-chemotherapy and at least 3 years after completion of chemotherapy
  Changes in self-reported peripheral neuropathy will be assessed using Functional Assessment of Cancer-Gynecology Oncology Group-Neurotoxicity (FACT/GOG-NTX-12), between pre-chemotherapy and at least 3 years after completion of chemotherapy in the Cohort B group (participants did not receive chemotherapy).
  FACT/GOG-NTX-12 is a questionnaire that includes 12 items inquiring about symptoms in the past 7 days (0=not at all to 4=very much) pertaining to numbness or tingling in hands/feet, discomfort in hands/feet, joint pain or muscle cramps, weakness all over, trouble hearing, ringing/buzzing in ears, buttoning buttons, trouble feeling the shape of small objects in hands, trouble walking, and pain in hands/feet in cold temperatures. The increasing score reflects worse neuropathy.
Changes in self-reported Fatigue-Cohort A | Pre-chemotherapy and at least 3 years after completion of chemotherapy
  Changes in self-reported Fatigue will be measured using Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) between pre-chemotherapy and at least 3 years after completion of chemotherapy in the Cohort A group (participants who received chemotherapy).
  Functional Assessment of Chronic Illness Therapy-Fatigue (TFACIT-F) is a 13-item scale that uses a 5-point Likert-type scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). The recall period is "during the past 7 days".
Changes in self-reported Fatigue-Cohort B | Pre-chemotherapy and at least 3 years after completion of chemotherapy
  Changes in self-reported Fatigue will be measured using Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) between pre-chemotherapy and at least 3 years after completion of chemotherapy in the Cohort B group (participants did not receive chemotherapy).
  Functional Assessment of Chronic Illness Therapy-Fatigue (TFACIT-F) is a 13-item scale that uses a 5-point Likert-type scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). The recall period is "during the past 7 days".

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Muss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials